CLINICAL TRIAL: NCT01547468
Title: Does Femoral Nerve Catheterization Reduce the Incidence of Post-Operative Delirium in Patients Presenting for Hip Fracture Repair?
Brief Title: A Comparison of Two Pain Control Techniques on Deliruim in Hip Fracture Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: inactivity and unable to complete due to manpower issues
Sponsor: Leslie Thomas (Other)
Collaborators: American Society of Anesthesiologists (Other)
Responsible Party: Sponsor-Investigator, Leslie Thomas, Anesthesiologist, Ochsner Health System
Organization: Ochsner Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010.198.C
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Hip Fracture
Keywords: hip fracture; elderly; delirium; broken hip; hip; surgery; orthopedic; orthopedic surgery; pain; anesthesia; Ochsner Clinic; Ochsner Hospital; Leslie Thomas MD; New Orleans; Louisiana
MeSH Terms: conditions — Hip Fractures; Delirium; Pain | interventions — Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous Opioids (Active Comparator)
  Interventions: Procedure: Intravenous Opioids
- Femoral Nerve Catheterization (Experimental)
  Interventions: Procedure: Femoral Nerve Catheterization

INTERVENTIONS:
Procedure: Femoral Nerve Catheterization — A femoral nerve catheter will be placed prior to surgery in this group.
  Other Names: FNC
  Arms: Femoral Nerve Catheterization
Procedure: Intravenous Opioids — Intravenous opioids will be given after surgery to provide pain relief to subjects assigned to this group.
  Other Names: IV opioids
  Arms: Intravenous Opioids

SUMMARY:
The purpose of this study is compare the rates of post-operative delirium between a group of people receiving intravenous (IV) pain control after hip fracture surgery and a group of people receiving a femoral nerve catheter for pain control. Post-operative delirium is confusion that can happen after the deep sleep of anesthesia. AThe hypothesis is that the group receiving the femoral nerve catheter for pain may have a lower incidence of delirium than the group receiveing IV pain medication.

DETAILED DESCRIPTION:
Subjects will have their hearing and vision tested. They will have their ability to think and analyze information tested using 4 questionnaires/ surveys: The Confusion Assesment Method (CAM), the Mini-Mental Status Examination (MMSE), Modified Blessed Dementia scale (MBDS), and Barthel's Activities of Daily Living (ADL). They will have pain medication prior to surgery based on the doctor's orders.

On the day of surgery, subjects will be randomized (like a flip of a coin) into one of two groups. One group will receive IV medication to control for pain after surgery. The other group will receive a femoral nerve catheter to control for pain after surgery.

A femoral nerve catheter is the small tubing that delivers numbing medicine to the nerves around the hips that control pain. This will be placed either before, during or soon after your surgery to help with pain after the surgery. This catheter is placed using an ultrasound machine. Subjects will still have pain medication through the IV before surgery if the catheter is put into their leg.

After surgery, you will be given the pain medication either through the IV or through the catheter in your leg. The catheter will be left in after surgery for 2-3 days delivering numbing medicine to the nerves. If subjects have the catheter in their leg and need more pain medication, the medication will be given to them through the IV.

Subjects will be visited by a member of the study staff on the second and third day after surgery. The study staff member will ask questions about the subject's ability to think and analyze information.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and older
* Presenting to Ochsner Main Campus with a hip fracture

Exclusion Criteria:

* Head trauma as reported in the medical record and/or patient response
* High impact fractures as reported in the medical record
* Aphasia as reported in the medical record and/or patient response
* Deafness, blindness as reported in the medical record and/or patient response
* True allergy (not sensitivity or side effects) to local anesthetics or opiates
* Pregnant
* Inability to complete study activities pre-operatively

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
number of participants developing delirium post-operatively | 3 days post-operatively

SECONDARY OUTCOMES:
the number of days admitted to the hospital post-operatively | participants will be followed for the duration of the hospital stay, an expected average of 4 days
Is there a difference in pain scores between subjects receiving the femoral nerve catheter vs. opioid only therapy for hip fracture pain using the visual analog scale (VAS) and consumption of pain medication for breakthrough pain relief? | post-op day 2 and again on post-op day 3
  Two VAS scores, at least 6 hours apart, will be taken from the medical chart on post-op day 2 and again on post-op day 3. The amount of pain medication (opioids), such as morphine, hydrocodone, oxycodone, etc. consumed will be recorded until discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Thomas, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States